CLINICAL TRIAL: NCT01134679
Title: Telephone Contacts to Improve Adherence to Dual Anti-Platelet Therapy Following Drug-Eluting Stent Implantation; A Randomized Controlled-Trial
Brief Title: (EASY)-IMProving Adherence to Clopidogrel Trial (IMPACT))
Acronym: EASY-IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Stéphane Rinfret, Professor under grant, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20424
Record Dates: First submitted 2009-07-23; First posted 2010-06-02 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stent; Clopidogrel; Aspirin
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phone calls (Experimental): Disease management with close patient follow-up, using phone calls.
  Interventions: Behavioral: Multi-disciplinary disease management approach

INTERVENTIONS:
Behavioral: Multi-disciplinary disease management approach — Follow up with phone calls

SUMMARY:
The purpose of this study is to test the impact of a multidisciplinary approach to improve the adhesion and persistence to Clopidogrel therapy. A simple and inexpensive therapy management involving a tighter monitoring of patients by nurses and pharmacists will improve the persistence and adhesion to Clopidogrel and Aspirin after the implantation of drug-eluting stents.

DETAILED DESCRIPTION:
Optimal treatment with Clopidogrel and Aspirin is critical for preventing complications after implantation of drug-eluting stents (DES). The premature cessation of Clopidogrel is a well recognized factor of thrombosis of stents, especially DES. Indeed, there remains a large portion of patients that prematurely stop clopidogrel. No study has demonstrated that a therapeutic management program could improve patient compliance to their antiplatelets. Through an open-label clinical study, two groups of patients who just received their DES will be compared: one with the usual protocol (consisting of seeing the cardiologist 6 weeks after the intervention) and one with the normal care supplemented by a simple and efficient follow-up (consisting of phone calls at 7 days, 1 month, 6 months and 9 months explaining the importance of antiplatelet therapy, evaluating the health of the patient and well received prescription from the pharmacy). Patients in both groups will receive a prescription to Clopidogrel and Aspirin (for 1 month), with 11 renewals.

ELIGIBILITY:
Inclusion Criteria:

* Percutaneous Coronary Intervention with implantation of Drug-Eluting Stent
* Prescription for Plavix and Aspirin

Exclusion Criteria:

* Patients frequenting more than one pharmacy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the number of days with available Clopidogrel and Aspirin (from pharmacy records) | 1 year

SECONDARY OUTCOMES:
the adhesion to Clopidogrel and Aspirin as self-reported by patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Rinfret, MD MSc, Principal Investigator — Fondation IUCPQ
Locations (1):
- Institut de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Rinfret S, Rodes-Cabau J, Bagur R, Dery JP, Dorais M, Larose E, Barbeau G, Gleeton O, Nguyen CM, Noel B, Proulx G, Roy L, Taillon I, De Larochelliere R, Bertrand OF; EASY-IMPACT Investigators. Telephone contact to improve adherence to dual antiplatelet therapy after drug-eluting stent implantation. Heart. 2013 Apr;99(8):562-9. doi: 10.1136/heartjnl-2012-303004. Epub 2013 Feb 23. PMID 23434769